CLINICAL TRIAL: NCT03587506
Title: The Relationship Between Periodic Limb Movement and Seizure Recurrence in Genetic Generalized Epilepsy
Brief Title: Periodic Limb Movement and Genetic Generalized Epilepsy
Acronym: Epilepsy
Status: Completed | Type: Observational
Sponsor: University of Alexandria (Other)
Responsible Party: Principal Investigator, Eman Hamdy, Assistant lecturer of Neurology, University of Alexandria
Other Study IDs: Alexandria Faculty of Medicine
Record Dates: First submitted 2018-07-01; First posted 2018-07-16 (Actual); Last update posted 2018-07-16 (Actual); Status verified 2018-07

CONDITIONS: Epilepsy Generalized Idiopathic Not Intractable
Keywords: Generalized epilepsy, idiopathic, periodic limb movement
MeSH Terms: conditions — Epilepsy, Generalized

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Patients: group: Group I (n=10) included patients who did not develop any major or minor seizure during the follow-up period and their follow up EEG was free of any epileptiform discharge
- Patients: group II: Group II (n=11) included patients who developed only minor seizures and their follow up EEG showed epileptiform discharge
- Patients: group III: Group III (n=9) were patients who developed one or more major seizures during the follow-up period whatever their EEG findings.
- Controls: healthy volunteers (n=30) who were not related to the patients and had no family history of epilepsy.

SUMMARY:
The study aimed to study the correlation between periodic limb movement occurring during sleep and the different parameters of genetic generalized epilepsy

DETAILED DESCRIPTION:
Although periodic limb movements are prevalent among patients with epilepsy, the exact relationship between these movements and epilepsy remains elusive. Objective: The aim of this work was to study the periodic limb movements among patients with genetic generalized epilepsy in relation to different clinical characteristics and seizure recurrence. Methods: Sixty individuals participated in this study: thirty of them were newly diagnosed with genetic generalized epilepsy and thirty were healthy individuals. Sleep quality was assessed using the Pittsburgh Sleep Quality Index questionnaire, and a standard polysomnographic study was conducted to all subjects. All patients then received sodium valproate in therapeutic doses and were followed up for six months. Electroencephalogram (EEG) was done after the follow-up period and seizure recurrence was assessed. Accordingly, patients were classified into three groups according to clinical seizure recurrence and follow-up EEG findings.

Periodic limb movement index and frequency were compared among the patients' groups and were correlated with different clinical characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed with genetic generalized epilepsy according to the ILAE 2010 criteria
* did not previously receive AEDs.
* The clinical seizures were either eyewitnessed by physicians or video-recorded to ensure they were true epileptic seizures.
* At least two unprovoked seizures occurring >24 hours apart

Exclusion Criteria:

* Patients with pre-existing psychiatric illnesses
* Patients with seizures due to toxic or metabolic causes (including glucose disturbance, uremia, and electrolytes disturbance), infections, or structural causes (such as neoplasms)
* Patients using hypnotic drugs

Ages: 9 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Thirty patients and thirty volunteer healthy controls were recruited. Patients were newly diagnosed with genetic generalized epilepsy according to the ILAE 2010 criteria who did not previously receive AEDs. The clinical seizures were either eye-witnessed by physicians or video-recorded to ensure they were true epileptic seizures. Age of participants ranged from 9 to 29 years. All patients recruited in this study had at least two unprovoked seizures occurring >24 hours apart. Patients with pre-existing psychiatric illnesses those with seizures due to toxic or metabolic causes ), infections, or structural causes, and those using hypnotic drugs were excluded. The control subjects were healthy volunteers who were not related to the patients and had no family history of epilepsy.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2015-09-03 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Seizure recurrence | 6 months
  Clinical major or minor seizure, and electrical seizure

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bazil CW. Sleep and Epilepsy. Semin Neurol. 2017 Aug;37(4):407-412. doi: 10.1055/s-0037-1604352. Epub 2017 Aug 24. No abstract available. PMID 28837987
- [Background] Malow BA, Fromes GA, Aldrich MS. Usefulness of polysomnography in epilepsy patients. Neurology. 1997 May;48(5):1389-94. doi: 10.1212/wnl.48.5.1389. PMID 9153478
- [Background] Yazdi Z, Sadeghniiat-Haghighi K, Naimian S, Zohal MA, Ghaniri M. Prevalence of Sleep Disorders and their Effects on Sleep Quality in Epileptic Patients. Basic Clin Neurosci. 2013 Winter;4(1):36-41. PMID 25337326
- [Background] Vetrugno R, D'Angelo R, Montagna P. Periodic limb movements in sleep and periodic limb movement disorder. Neurol Sci. 2007 Jan;28 Suppl 1:S9-S14. doi: 10.1007/s10072-007-0733-0. No abstract available. PMID 17235435
- [Background] Karadeniz D, Ondze B, Besset A, Billiard M. EEG arousals and awakenings in relation with periodic leg movements during sleep. J Sleep Res. 2000 Sep;9(3):273-7. doi: 10.1046/j.1365-2869.2000.00202.x. PMID 11012867
- [Background] Parrino L, Ferri R, Bruni O, Terzano MG. Cyclic alternating pattern (CAP): the marker of sleep instability. Sleep Med Rev. 2012 Feb;16(1):27-45. doi: 10.1016/j.smrv.2011.02.003. Epub 2011 May 26. PMID 21616693
- [Background] Allena M, Campus C, Morrone E, De Carli F, Garbarino S, Manfredi C, Sebastiano DR, Ferrillo F. Periodic limb movements both in non-REM and REM sleep: relationships between cerebral and autonomic activities. Clin Neurophysiol. 2009 Jul;120(7):1282-90. doi: 10.1016/j.clinph.2009.04.021. Epub 2009 Jun 7. PMID 19505849
- [Background] Berg AT, Millichap JJ. The 2010 revised classification of seizures and epilepsy. Continuum (Minneap Minn). 2013 Jun;19(3 Epilepsy):571-97. doi: 10.1212/01.CON.0000431377.44312.9e. PMID 23739099
- [Background] Fisher RS, Acevedo C, Arzimanoglou A, Bogacz A, Cross JH, Elger CE, Engel J Jr, Forsgren L, French JA, Glynn M, Hesdorffer DC, Lee BI, Mathern GW, Moshe SL, Perucca E, Scheffer IE, Tomson T, Watanabe M, Wiebe S. ILAE official report: a practical clinical definition of epilepsy. Epilepsia. 2014 Apr;55(4):475-82. doi: 10.1111/epi.12550. Epub 2014 Apr 14. PMID 24730690
- [Background] Jagannath A, Peirson SN, Foster RG. Sleep and circadian rhythm disruption in neuropsychiatric illness. Curr Opin Neurobiol. 2013 Oct;23(5):888-94. doi: 10.1016/j.conb.2013.03.008. Epub 2013 Apr 23. PMID 23618559
- [Background] Flink R, Pedersen B, Guekht AB, Malmgren K, Michelucci R, Neville B, Pinto F, Stephani U, Ozkara C; Commission of European Affairs of the International League Against Epilepsy: Subcommission on European Guidelines. Guidelines for the use of EEG methodology in the diagnosis of epilepsy. International League Against Epilepsy: commission report. Commission on European Affairs: Subcommission on European Guidelines. Acta Neurol Scand. 2002 Jul;106(1):1-7. doi: 10.1034/j.1600-0404.2002.01361.x. PMID 12067321
- [Background] Glauser T, Ben-Menachem E, Bourgeois B, Cnaan A, Guerreiro C, Kalviainen R, Mattson R, French JA, Perucca E, Tomson T; ILAE Subcommission on AED Guidelines. Updated ILAE evidence review of antiepileptic drug efficacy and effectiveness as initial monotherapy for epileptic seizures and syndromes. Epilepsia. 2013 Mar;54(3):551-63. doi: 10.1111/epi.12074. Epub 2013 Jan 25. PMID 23350722
- [Background] Khatami R, Zutter D, Siegel A, Mathis J, Donati F, Bassetti CL. Sleep-wake habits and disorders in a series of 100 adult epilepsy patients--a prospective study. Seizure. 2006 Jul;15(5):299-306. doi: 10.1016/j.seizure.2006.02.018. Epub 2006 Mar 20. PMID 16546407
- [Background] Parrino L, Boselli M, Buccino GP, Spaggiari MC, Di Giovanni G, Terzano MG. The cyclic alternating pattern plays a gate-control on periodic limb movements during non-rapid eye movement sleep. J Clin Neurophysiol. 1996 Jul;13(4):314-23. doi: 10.1097/00004691-199607000-00005. PMID 8858493
- [Background] Parrino L, Smerieri A, Spaggiari MC, Terzano MG. Cyclic alternating pattern (CAP) and epilepsy during sleep: how a physiological rhythm modulates a pathological event. Clin Neurophysiol. 2000 Sep;111 Suppl 2:S39-46. doi: 10.1016/s1388-2457(00)00400-4. PMID 10996553